CLINICAL TRIAL: NCT00211120
Title: Correction of Hemoglobin and Outcomes In Renal Insufficiency
Brief Title: Correction of Hemoglobin and Outcomes in Renal Insufficiency (CHOIR)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped by the DSMB due to a trend toward more adverse events in the higher hemoglobin (Hb) arm and <5% chance that the study would show benefit for higher Hb.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004588
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-03

CONDITIONS: Anemia
Keywords: Anemia; Low Blood Count; Chronic Kidney Failure; Chronic Kidney Disease
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The purpose of this study is to compare the outcomes of patients with chronic kidney disease (CKD) randomly assigned to 2 treatment groups, which differ only in their targeted hemoglobin levels. This study will test the primary hypothesis that the level of anemia correction with once weekly dosing of PROCRITÂ® (Epoetin alfa) in patients with chronic kidney disease will decrease mortality and cardiovascular morbidity.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized, multi-center study in patients with CKD. Patients who meet the selection criteria will be randomly assigned to one of two treatment arms: GROUP A: PROCRIT® (Epoetin alfa) therapy directed at maintaining the hemoglobin level as close to 13.5 g/dL as possible (may be slightly higher or lower) or GROUP B: PROCRIT® (Epoetin alfa) therapy directed at maintaining the hemoglobin level as close to 11.3 g/dL as possible (may be slightly higher or lower).

Patients will receive weekly doses of PROCRIT® (Epoetin alfa). Subsequent doses of PROCRIT® will be given weekly as needed with dose adjustments made to maintain the hemoglobin (Hb) as close to the target level as possible until the initiation of Renal Replacement Therapy (RRT) or 36 months, whichever comes first.

The purpose of this study is to compare the outcomes of patients with CKD randomly assigned to 2 treatment groups, which differ only in their targeted hemoglobin levels. This study will test the primary hypothesis that the level of anemia correction with once weekly dosing of PROCRIT® (Epoetin alfa) in patients with chronic kidney disease will decrease mortality and cardiovascular morbidity. Patients will receive a starting dose of PROCRIT® 10,000 Units (U) subcutaneously (SC) 1x / week. After 3 weekly doses, subsequent doses and dosing intervals of PROCRIT®, up to a maximum dose of 20,000 U for 36 months, will be adjusted based on an assessment of the two most recent hemoglobin values.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease:Glomerular filtration rate (GFR) > 15 mL/min and > 50 mL/min as calculated by the central lab. HB<11 g/dL upon study enrollment. The GFR for assessment of patient eligibility will be determined using the formula derived from the Modification of Diet for Renal Disease (MDRD) Study.

Exclusion Criteria:

* Pregnant or lactating women
* Presence of uncontrolled hypertension
* Known hypersensitivity to mammalian cell-derived products or human albumin
* Active gastrointestinal bleeding
* Iron overload defined as a transferrin saturation >70% or ferritin >1000 ng/mL
* History of frequent blood transfusions in the past 6 months
* Unstable angina or angina pectoris at rest
* Severe chronic obstructive pulmonary disease requiring routine use of supplemental oxygen
* Severe liver dysfunction that is defined by an international normalized ratio >2.0, not caused by an anticoagulant
* Severe malnutrition
* Active hematological disease (eg, sickle cell anemia, thalassemia)
* Active malignancy (usually defined as malignancy requiring current chemotherapy or radiotherapy)
* Patients with current seizure disorder or activity
* Patients currently receiving RRT (patient can not be on dialysis or have had a kidney transplant)
* Patients who have received Epoetin Alpha within 6 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1432 (Actual)
Dates: Start 2002-03; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be a composite consisting of mortality (all cause), myocardial infarction, stroke, and CHF hospitalization (not including those hospitalizations during which RRT occurs)

SECONDARY OUTCOMES:
All cause mortality; Myocardial infarction; Stroke; RRT;CHF, Cardiovascular and all cause hospitalizations, Change from baseline in hemoglobin, Quality of Life Scores (SF36, KDQ, LASA), transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Singh AK, Szczech L, Tang KL, Barnhart H, Sapp S, Wolfson M, Reddan D; CHOIR Investigators. Correction of anemia with epoetin alfa in chronic kidney disease. N Engl J Med. 2006 Nov 16;355(20):2085-98. doi: 10.1056/NEJMoa065485. PMID 17108343
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: Correction of Hemoglobin and Outcomes in Renal Insufficiency (CHOIR)) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=600&filename=CR004588_CSR.pdf